CLINICAL TRIAL: NCT01258647
Title: Caterpillar Cereal: Maternal and Infant Acceptability
Brief Title: Acceptability of a Cereal for Complementary Feeding of Infants and Young Children Made From Caterpillars
Acronym: CAT01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Kinshasa School of Public Health (Other); University of California, Davis (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Carl Bose, Prinicipal Investigator, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10-0509
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Malnutrition; Stunting of Growth
Keywords: infant nutrition; complementary feeding; malnutrition; stunting of growth
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Feeding group (Experimental): The feeding group will include 20 mother/infant dyads. The infants will be between 8 and 10 months of age.
  Interventions: Dietary Supplement: caterpillar cereal

INTERVENTIONS:
Dietary Supplement: caterpillar cereal — A 30 gram portion of a cereal containing one part dried, ground caterpillar, one part corn flour and small quantities of sugar and palm oil will be evaluated by the mothers and then fed daily for seven days to infants.

SUMMARY:
Two in every three infants in rural areas of the Democratic Republic of Congo (DRC) suffer from stunting of linear growth by 12 months of age. Stunting presumably results from breast milk supplementation after 6 months of age with complementary foods (CF) that provide inadequate protein and micronutrients. Although supplementation with selected micronutrients may avoid certain deficiency states, CF with animal source foods may be necessary to avoid stunting. Meat is not readily available in many Central African countries. However caterpillars, which are locally available and abundant, are a common staple in adult diets and may be a suitable substitute for animal source proteins in CF. The investigators developed a cereal made from dried caterpillars that has a nutrient content that appears to be ideal for CF. Maternal and infant acceptability will be evaluated in 20 mothers and their 8 month old infants. The investigators hypothesize that this cereal will be accepted by both mothers and infants: acceptability will be based on a priori definitions.

DETAILED DESCRIPTION:
In preparation for a controlled study of the efficacy of daily intake of caterpillar cereal versus the usual diet from 6 to 18 months of age in reducing the rate of stunting of linear growth, and the improvement in other health outcomes, we will conduct an acceptability trial. In this trial, we will test the mothers' acceptance of the caterpillar cereal and their willingness to feed their young children this product. We will also test the infants' acceptance and their capacity to consume quantities required in the controlled trial necessary to deliver the desired quantities of micronutrients.

Study Design

A cohort of 20 mother-infant dyads will be recruited. The site of recruitment will be the area Health Center. Infants will be between 8 and 10 months of age and will have no major health problems. Infants with minor, inter-current illnesses at the time of recruitment that might interfere with oral intake will be excluded. After informed consent, maternal and infant acceptability will be tested using the methods described below.

Maternal Acceptability

Mothers will be provided with a 30 g portion of caterpillar cereal and will be instructed in the proper technique for preparation. After preparation, mothers will be asked to evaluate five features of the cereal. They will also be asked to provide their overall impression of the cereal. In each category, the evaluation will be assigned a numerical score using a five-part Likert scale, from "like very much" to "dislike very much".

The evaluation will be conducted by the Community Coordinator (CC) who will provide instruction about cereal preparation and administer the evaluative tool. Each evaluation will be conducted confidentially. Mothers will not be aware of the response of other mothers. At the conclusion of a one-week period of feeding (see below), a questionnaire will be administered to assess mothers' attitudes about their willingness to participate in a one-year study of cereal feeding.

We do not intend to evaluate their attitudes about food preparation. The recommended preparation technique of the caterpillar cereal is very similar to preparation of enriched soy cereal in our ongoing complementary feeding study. This involves boiling water and cooking the cereal for approximately three minutes. Although this preparation technique is burdensome, it has not compromised compliance in the ongoing study. Therefore, we would expect a similar response from mothers in the proposed study.

Infant Acceptability

Following the evaluation of maternal acceptability, each mother will be provided with a one-week supply of caterpillar cereal (7 individual packets containing 30 g each). She will be instructed to begin daily feedings on the following day, and to continue until the cereal packets have all been used. The first feeding will occur during a home visit by the CC, who will repeat the preparation instructions, and will observe the first feeding. The CC will return to the home on alternate days throughout the week to reinforce instructions regarding preparation, and to make observations about infant feeding habits. Although frequent visits may influence the likelihood of maternal compliance and hence may mislead investigators about maternal acceptability, it will not effect infant acceptability.

Mothers will be instructed not to feed the cereal to other household members, and will be asked to return uneaten cereal to the original packet for collection by the CC at the end of the week.

On the 8th day, the day following the completion of use of the cereal, the CC will return to the home for the purpose of data collection. The CC will administer a 24-hour dietary recall, and collect all cereal packets. In addition, mothers will be asked questions about the infant's health status.

ELIGIBILITY:
Inclusion Criteria:

* Any mother-infant dyad living within each a study community in the Equateur Province. Infants must be 8-10 months of age at the time of recruitment.

Exclusion Criteria:

* Infants with minor inter-current illness that may interfere with oral intake
* Infants of multiple gestation births
* Infants with congenital anomalies
* Infants likely to receive free or subsidized complementary foods (or infant formula)

Ages: 8 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Maternal acceptability | Maternal acceptability will be measured on the first day of the trial.
  Maternal acceptability will be defined as a median score for each of 5 features (smell, taste, texture, color, consistency, overall impression) of 3 or greater on a 5 point Likert scale.
Infant acceptability | Infant acceptability will be measured during the one week study period.
  Each mother will be provided with a one-week supply of caterpillar cereal and will be instructed to begin daily feedings for a period of one week. Infant acceptability will be defined as the consumption of greater than 75% of the total cereal allotment by all infants during the last four days of feeding.

SECONDARY OUTCOMES:
Infant tolerance | This outcome will be measured throughout the one week intervention.
  During the visits by the Community Coordinator, mothers will be asked question about the infant's health status and specifically about any signs or symptoms attributable to feeding.
  Tolerance will be defined as the absence of signs or symptoms attributable to cereal consumption (diarrhea or emesis unless other family members have developed these symptoms during the week of feeding).

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Bose, MD, Principal Investigator — University of North Carolina
Locations (1):
- Kinshasa School of Public Health, Kinshasa, Republic of the Congo